CLINICAL TRIAL: NCT05188521
Title: Baricitinib (LY3009104) in the Treatment of Cutaneous Lichen Planus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aaron R. Mangold (Other)
Responsible Party: Sponsor-Investigator, Aaron R. Mangold, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-003075
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Cutaneous Lichen Planus
MeSH Terms: conditions — Lichen Planus | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cutaneous LP (Experimental): Subjects with a diagnosis of cutaneous LP will receive Baricitinib (LY3009104) for a 16 weeks treatment period
  Interventions: Drug: Baricitinib (LY3009104) 2 mg
- Dose Escalation Extension Group (Experimental): Subject that demonstrate a response to the 16 weeks of treatment with 2 mg of Baricitinib (LY3009104), but have not achieved a PGA 0 will receive 4 mg of Baricitinib (LY3009104) for 12 weeks
  Interventions: Drug: Baricitinib (LY3009104) 4 mg

INTERVENTIONS:
Drug: Baricitinib (LY3009104) 2 mg — 2 mg orally administered once daily for 16 weeks
  Arms: Cutaneous LP
Drug: Baricitinib (LY3009104) 4 mg — 4 mg orally administered once daily for 12 weeks
  Arms: Dose Escalation Extension Group

SUMMARY:
This research study is evaluating the safety and efficacy of Baricitinib in treating Cutaneous Lichen Planus (LP).

ELIGIBILITY:
Inclusion Criteria

* Subjects must be able to understand and comply with the requirements of the study and communicate with the investigator. Subjects must give written, signed, and dated informed consent before any study related activity is performed. When appropriate, a legal representative will sign the informed consent according to local laws and regulation
* Both men and women must be at least 18 years of age at the time of screening
* Subjects must have clinical and histological features of LP
* LP requiring systemic treatment
* Subjects must have treatment naïve cutaneous LP or treatment refractory disease, as defined by failure of at least one established treatment for LP. Failure of prior therapy: topical treatment, systemic immunosuppressant, oral metronidazole, oral sulfasalazine, oral retinoid

Exclusion Criteria

* On excluded therapies, not on a stable dose of a therapy, or incompletely washed out for a therapy
* Known hypersensitivity or other adverse reaction to Baricitinib (LY3009104)
* Variants of LP deemed by the investigators to be inappropriate for Baricitinib (LY3009104) including but not limited to:

  o Drug-induced LP: Predominant non-cutaneous variants of LP, note that individuals can have disease in non-cutaneous areas; however, they must also have cutaneous disease Lichen Planopilaris or Oral Lichen planus
* Pregnant or nursing (lactating) women (pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test)
* Women of childbearing potential [Post-menopausal or not of child-bearing potential is defined by 1 year of natural (spontaneous) amenorrhea or surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least 6 weeks ago. Oophorectomy alone must be confirmed by follow up hormone level assessment to be considered not of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using basic methods of contraception which includes:

  * Total abstinence (Periodic abstinence and withdrawal are not acceptable methods of contraception)
  * Female sterilization (bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks before taking study treatment. Oophorectomy alone requires follow up hormone level assessment for fertility.
  * Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject.
  * Barrier methods of contraception: condom or occlusive cap.
  * Use of oral, injected or implanted hormonal methods of contraception or other forms or hormonal contraception that have complete efficacy (failure <1%). (The dose of the contraceptive should be stable for 3 months)
* Active ongoing inflammatory diseases of the skin other than LP that might confound the evaluation of the benefit of Baricitinib (LY3009104)
* Underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal conditions) which, in the opinion of the investigator, significantly immunocompromises the subject and/or places the subject at unacceptable risk for receiving an immunomodulatory therapy
* Moderate-to-severe renal impairment including patients with estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m^2
* Active systemic infections during the 2 weeks prior to randomization (common cold viruses excluded) or any infection that reoccurs on a regular basis
* Current severe progressive or uncontrolled disease which the investigator renders the subject unsuitable for the trial or puts the subject at increased risk
* Have had any major surgery within 8 weeks prior to screening or will require major surgery during the study that, in the opinion of the investigator would pose an unacceptable risk to the patient.
* Have experienced any of the following within 12 weeks of screening: VTE (DVT/pulmonary embolism [PE]), myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure.
* Have a history of recurrent (≥ 2) VTE (DVT/PE).
* Have a history of lymphoproliferative disease; have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; have active primary or recurrent malignant disease; or have been in remission from clinically significant malignancy for <5 years prior to randomization.
* Have had symptomatic herpes zoster infection within 12 weeks prior to randomization.
* Have a history of disseminated/complicated herpes zoster (for example, ophthalmic zoster or CNS involvement).
* ALT or AST >2 x upper limits of normal (ULN); alkaline phosphatase (ALP) ≥2 x ULN; total bilirubin ≥1.5 x ULN; hemoglobin <10 g/dL (100.0 g/L); total white blood cell count <3000 cells/μL (<3.00 x 103/μL or <3.00 billion/L); neutropenia (absolute neutrophil count [ANC] <1500 cells/μL) (<1.50 x 103/μL or <1.50 billion/L); lymphopenia (lymphocyte count <1000 cells/μL) (<1.00 x 103/μL or <1.00 billion/L); thrombocytopenia (platelets <100,000 cells/μL) (<100 x 103/μL or <100 billion/L) Note: Patients who are HBcAb-positive and HBV DNA-negative may be enrolled in the study but will require additional HBV DNA monitoring during the study.
* Have a positive test for hepatitis B virus (HBV) defined as positive for hepatitis B surface antigen (HBsAg), or positive for hepatitis B core antibody (HBcAb) and positive for hepatitis B virus deoxyribonucleic acid (HBV DNA). Note: Patients who are HBcAb-positive and HBV DNA-negative may be enrolled in the study but will require additional HBV DNA monitoring during the study.
* Have hepatitis C virus (HCV) infection (hepatitis C antibody-positive and HCV ribonucleic acid [RNA]-positive).

Note: Patients who have documented anti-HCV treatment for a past HCV infection AND are HCV RNA-negative may be enrolled in the study.

* Have evidence of HIV infection and/or positive HIV antibodies.
* Have had household contact with a person with active TB and did not receive appropriate and documented prophylaxis for TB.
* Have evidence of active TB or latent TB
* Have evidence of active TB, defined in this study as the following:

  * Positive purified protein derivative (PPD) test (≥5 mm induration between approximately 2 and 3 days after application, regardless of vaccination history), medical history, clinical features, and abnormal chest x-ray at screening.
  * QuantiFERON®-TB Gold test or T-SPOT®.TB test (as available and if compliant with local TB guidelines) may be used instead of the PPD test. Patients are excluded from the study if the test is not negative and there is clinical evidence of active TB. Exception: patients with a history of active TB who have documented evidence of appropriate treatment, have no history of re-exposure since their treatment was completed, have no clinical features of active TB, and have a screening chest x-ray with no evidence of active TB may be enrolled if other entry criteria met. Such patients would not be required to undergo the protocol-specific TB testing for PPD, QuantiFERON®-TB Gold test, or T-SPOT®.TB test but must have a chest x-ray at screening (i.e., chest imaging performed within the past 6 months will not be accepted).
* Have evidence of untreated/inadequately or inappropriately treated latent TB, defined in this study as the following:

  * Positive PPD test, no clinical features consistent with active TB, and a chest x-ray with no evidence of active TB at screening; or
  * If the PPD test is positive and the patient has no medical history or chest x-ray findings consistent with active TB, the patient may have a QuantiFERON®-TB Gold test or T-SPOT®.TB test (as available and if compliant with local TB guidelines). If the test results are not negative, the patient will be considered to have latent TB (for purposes of this study); or
  * QuantiFERON®-TB Gold test or T- SPOT®.TB test (as available and if compliant with local TB guidelines) may be used instead of the PPD test. If the test results are positive, the patient will be considered to have latent TB. If the test is not negative, the test may be repeated once within approximately 2 weeks of the initial value. If the repeat test results are again not negative, the patient will be considered to have latent TB (for purposes of this study).
* Have been exposed to a live vaccine within 12 weeks of randomization or are expected to need/receive a live vaccine during the course of the study (with the exception of herpes zoster vaccination).
* Have donated more than a single unit of blood within 4 weeks prior to screening or intend to donate blood during the course of the study.
* Have a history of intravenous drug abuse, other illicit drug abuse, or chronic alcohol abuse within the 2 years prior to screening or are concurrently using, or expected to use during the study, illicit drugs (including marijuana).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron R Mangold, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- [Derived] Zhang N, Stockard AL, Leibovit-Reiben Z, Hwang AS, Kechter JA, Brumfiel CM, Patel MH, Bhullar P, Morken C, Boudreaux BW, Nassir S, Yousif M, Ogbaudu E, Xie F, Zunich S, Branch E, Dueck A, Lehman J, Pittelkow MR, Mangold AR. Repurposing the composite assessment of index lesion severity scoring system in cutaneous lichen planus. Arch Dermatol Res. 2025 Feb 14;317(1):413. doi: 10.1007/s00403-025-03996-4. PMID 39951132
- [Derived] Hwang A, Kechter J, Do T, Hughes A, Zhang N, Li X, Wasikowski R, Brumfiel C, Patel M, Boudreaux B, Bhullar P, Nassir S, Yousif M, DiCaudo DJ, Fox J, Gharaee-Kermani M, Xing X, Zunich S, Branch E, Kahlenberg JM, Billi AC, Plazyo O, Tsoi LC, Pittelkow MR, Gudjonsson JE, Mangold AR. Oral Baricitinib in the Treatment of Cutaneous Lichen Planus. medRxiv [Preprint]. 2024 Jan 11:2024.01.09.24300946. doi: 10.1101/2024.01.09.24300946. PMID 38260663

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 11 participants that concluded the initial 16 weeks of treatment, six were eligible to enroll in the dose escalation extension for an additional 12 weeks of treatment. Five of the six elected to continue with the study.
Period: Baricitinib 2mg Initial Study
Arm/Group | Cutaneous LP | Dose Escalation Extension Group
Started | 12 | 0
Completed | 11 | 0
Not Completed | 1 | 0
Not completed — Travel issues | 1 | 0
Period: Baricitinib 4mg Extension Study
Arm/Group | Cutaneous LP | Dose Escalation Extension Group
Started | 0 | 5
Completed | 0 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of twelve participants were enrolled in the overall study, which contained a dose escalation extension. Five of the twelve completed the dose escalation extension, resulting in a total of seventeen participants analyzed for the Baseline Measures overall.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cutaneous LP | Dose Escalation Extension Group | Total
Number analyzed (Participants) | 12 | 5 | 17
Age, Categorical [Count of Participants; unit: Participants] — Population: Data collected from each group are being reported separately to avoid multi-counted participants.
  Participants
    Baricitinib 2mg Initial Study: number analyzed (Participants) | 12 | 0 | 12
    Baricitinib 2mg Initial Study: <=18 years | 0 |  | 0
    Baricitinib 2mg Initial Study: Between 18 and 65 years | 5 |  | 5
    Baricitinib 2mg Initial Study: >=65 years | 7 |  | 7
    Baricitinib 4mg Extension Study: number analyzed (Participants) | 0 | 5 | 5
    Baricitinib 4mg Extension Study: <=18 years |  | 0 | 0
    Baricitinib 4mg Extension Study: Between 18 and 65 years |  | 3 | 3
    Baricitinib 4mg Extension Study: >=65 years |  | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data collected from each study are being reported separately to avoid multi-counted participants.
  Participants
    Baricitinib 2mg Initial Study: number analyzed (Participants) | 12 | 0 | 12
    Baricitinib 2mg Initial Study: Female | 11 |  | 11
    Baricitinib 2mg Initial Study: Male | 1 |  | 1
    Baricitinib 4mg Extension Study: number analyzed (Participants) | 0 | 5 | 5
    Baricitinib 4mg Extension Study: Female |  | 5 | 5
    Baricitinib 4mg Extension Study: Male |  | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data collected from each study are being reported separately to avoid multi-counted participants.
  Participants
    Baricitinib 2mg Initial Study: number analyzed (Participants) | 12 | 0 | 12
    Baricitinib 2mg Initial Study: Hispanic or Latino | 2 |  | 2
    Baricitinib 2mg Initial Study: Not Hispanic or Latino | 10 |  | 10
    Baricitinib 2mg Initial Study: Unknown or Not Reported | 0 |  | 0
    Baricitinib 4mg Extension Study: number analyzed (Participants) | 0 | 5 | 5
    Baricitinib 4mg Extension Study: Hispanic or Latino |  | 1 | 1
    Baricitinib 4mg Extension Study: Not Hispanic or Latino |  | 4 | 4
    Baricitinib 4mg Extension Study: Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data collected from each study are being reported separately to avoid multi-counted participants.
  Participants
    Baricitinib 2mg Initial Study: number analyzed (Participants) | 12 | 0 | 12
    Baricitinib 2mg Initial Study: American Indian or Alaska Native | 0 |  | 0
    Baricitinib 2mg Initial Study: Asian | 0 |  | 0
    Baricitinib 2mg Initial Study: Native Hawaiian or Other Pacific Islander | 0 |  | 0
    Baricitinib 2mg Initial Study: Black or African American | 1 |  | 1
    Baricitinib 2mg Initial Study: White | 9 |  | 9
    Baricitinib 2mg Initial Study: More than one race | 0 |  | 0
    Baricitinib 2mg Initial Study: Unknown or Not Reported | 2 |  | 2
    Baricitinib 4mg Extension Study: number analyzed (Participants) | 0 | 5 | 5
    Baricitinib 4mg Extension Study: American Indian or Alaska Native |  | 0 | 0
    Baricitinib 4mg Extension Study: Asian |  | 0 | 0
    Baricitinib 4mg Extension Study: Native Hawaiian or Other Pacific Islander |  | 0 | 0
    Baricitinib 4mg Extension Study: Black or African American |  | 0 | 0
    Baricitinib 4mg Extension Study: White |  | 4 | 4
    Baricitinib 4mg Extension Study: More than one race |  | 0 | 0
    Baricitinib 4mg Extension Study: Unknown or Not Reported |  | 1 | 1
Region of Enrollment [Number; unit: participants] — Baricitinib 2mg Initial Study Population: Data collected from each study are being reported separately to avoid multi-counted participants.
  participants
    United States: number analyzed (Participants) | 12 | 0 | 12
    United States | 12 |  | 12
Region of Enrollment [Number; unit: participants] — Baricitinib 4mg Extension Study Population: Data collected from each study are being reported separately to avoid multi-counted participants.
  participants
    United States: number analyzed (Participants) | 0 | 5 | 5
    United States |  | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Physician Global Assessment (PGA) of Skin Overall Response
Description: Measured by Physician Global Assessment (PGA) of skin by grade. The assessment ranges from Grade 0 (completely clear with no evidence of disease; 100% improvement) to Grade 6 (worse than at baseline evaluation by ≥25%; more progressive disease).
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Cutaneous LP
Number analyzed (Participants) | 11
Participants
  Grade 0 | 5
  Grade 1 | 5
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 1
  Grade 5 | 0
  Grade 6 | 0

2. Secondary Outcome: Change in Modified CAILS Score of the Cutaneous Index Treatment
Description: Measured by Modified CAILS-Clinical Assessment Scale of Severity for Index Lesion Signs and Symptoms (mCAILS). The area of the lesion is measured with digital planimetry. Lesion size by square centimeter is graded on a scale of 0 to 18, where 0 is no measurable area and 18 is greater than 300 centimeters. The higher the score the larger the lesion.
Time Frame: Baseline, Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cutaneous LP
Number analyzed (Participants) | 12
score on a scale | -10.6 (2.9)
Statistical Analysis 1: Comparison: Cutaneous LP; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Modified CAILS Score of the Cutaneous Index Treatment
Description: as for outcome 2
Time Frame: Week 16, Week 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose Escalation Extension Group
Number analyzed (Participants) | 5
score on a scale | -1.1 (4.3)
Statistical Analysis 1: Comparison: Dose Escalation Extension Group; Test type: Superiority; p = 0.593, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Skin Lesion Count
Description: Change in the number of subject's skin lesions from baseline to Week 16.
Time Frame: Baseline, Week 16
Measure: Mean (Standard Deviation); unit: number of skin lesions
Arm/Group | Cutaneous LP
Number analyzed (Participants) | 12
number of skin lesions | -134.8 (157.0)
Statistical Analysis 1: Comparison: Cutaneous LP; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Skin Lesion Count
Description: Change in the number of subject's skin lesions from Week 16 to Week 28.
Time Frame: Week 16, Week 28
Measure: Mean (Standard Deviation); unit: number of skin lesions
Arm/Group | Dose Escalation Extension Group
Number analyzed (Participants) | 5
number of skin lesions | -12.6 (17.6)
Statistical Analysis 1: Comparison: Dose Escalation Extension Group; Test type: Superiority; p = 0.138, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Pruritus Numerical Rating Scale (NRS)
Description: The Pruritus NRS is self-reported single question that asks "how severe itching has been over the last 24 hours". The response uses a scale of 0 (no itching) to 10 (severe itching). The higher the score, the worse the itching.
Time Frame: Baseline, Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cutaneous LP
Number analyzed (Participants) | 11
score on a scale | -5.3 (2.6)
Statistical Analysis 1: Comparison: Cutaneous LP; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in Pruritus Numerical Rating Scale (NRS)
Description: as for outcome 6
Time Frame: Week 16, Week 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose Escalation Extension Group
Number analyzed (Participants) | 5
score on a scale | -1.0 (2.2)
Statistical Analysis 1: Comparison: Dose Escalation Extension Group; Test type: Superiority; p = 0.357, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change in Overall Skindex-16 Assessment
Description: This validated questionnaire is a 16-item, participant-reported survey used to assess quality of life impacts due to the participant's skin condition. Scores range from 0 to 6, where 0 is never bothered by the skin condition and 6 is always bothered by the skin condition. Results are summed to produce an overall score, ranging from 0 to 96, where lower scores indicated a higher level of quality of life.
Time Frame: Baseline, Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cutaneous LP
Number analyzed (Participants) | 12
score on a scale | -37.3 (18.3)
Statistical Analysis 1: Comparison: Cutaneous LP; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Overall Skindex-16 Assessment
Description: as for outcome 8
Time Frame: Week 16, Week 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose Escalation Extension Group
Number analyzed (Participants) | 5
score on a scale | 4.0 (12.3)
Statistical Analysis 1: Comparison: Dose Escalation Extension Group; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant from baseline to 30 days following the last administration of the study product. The Baricitinib 2mg group was followed for a total of approximately 5 months. The participants who continued in the Baricitinib 4mg extension group were followed for a total of approximately 9 months.
Arm/Group | Cutaneous LP | Dose Escalation Extension Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/5
Other Adverse Events (participants affected / at risk) | 8/12 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cutaneous LP (N=12) | Dose Escalation Extension Group (N=5)
Hospitalization due to fall (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cutaneous LP (N=12) | Dose Escalation Extension Group (N=5)
Foot/leg pain/cramps (General disorders) | 2 (2) | 1 (1)
Headache (General disorders) | 2 (2) | 0 (0)
Constipation (General disorders) | 0 (0) | 1 (2)
Night Sweats (General disorders) | 0 (0) | 1 (1)
Cold symptoms (General disorders) | 1 (1) | 1 (1)
COVID-19 (General disorders) | 1 (1) | 0 (0)
Subconjunctival hemorrhage in left eye (General disorders) | 1 (1) | 0 (0)
Chest pain/tenderness (General disorders) | 1 (2) | 0 (0)
Hives (General disorders) | 1 (1) | 0 (0)
Ankle swelling (General disorders) | 1 (1) | 0 (0)
Rash on chest/back (General disorders) | 1 (1) | 0 (0)
Side pain (General disorders) | 0 (0) | 1 (1)
Visual field changes (General disorders) | 0 (0) | 1 (1)
Lichen planus flare (General disorders) | 1 (1) | 0 (0)
Low neutrophil count (General disorders) | 1 (1) | 0 (0)
Elevated creatine kinase (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT05188521/Prot_SAP_000.pdf